CLINICAL TRIAL: NCT05849012
Title: A Pilot Study Examining Low Sulfur Diet as Treatment for Persistent Symptoms in Quiescent Crohn's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Allen Lee, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00218796
Record Dates: First submitted 2023-04-25; First posted 2023-05-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease in Remission
Keywords: Crohn's disease; Quiescent Crohn's disease; Low sulfur diet; Microbiome
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: 20 subjects will be randomized to receive either a low sulfur diet or usual diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Sulfur Diet (Experimental): Participants in this group will follow a low sulfur diet. This diet decreases the amount of animal products (including meat, dairy, and eggs) as well as sulfur additives in the diet. The main types of foods in the low sulfur diet include fruits, vegetables, whole grains, nuts, seeds, and soy products.
  Interventions: Other: Low Sulfur Diet
- Usual Diet (Active Comparator): Participants in this group will follow a standard of care usual diet for 8 weeks.
  Interventions: Other: Usual Diet

INTERVENTIONS:
Other: Low Sulfur Diet — Subjects will be placed on a low sulfur diet for 8 weeks with the support of a nutritionist.
  In addition, participants will be asked to complete: surveys, lactulose-mannitol test, glucose hydrogen breath test, blood samples, visceral sensation test, 24-hour urine sample for sulfate level, provide stool samples, optional colonoscopy.
  Arms: Low Sulfur Diet
Other: Usual Diet — Subjects will continue on their usual diet for 8 weeks. At the end of 8 weeks, if participants are interested, they will be offered treatment with low sulfur diet for 8 weeks with the support of a nutritionist.
  In addition, participants will be asked to complete: surveys, lactulose-mannitol test, glucose hydrogen breath test, blood samples, visceral sensation test, 24-hour urine sample for sulfate level, provide stool samples, optional colonoscopy.
  Arms: Usual Diet

SUMMARY:
The goal of this study is to learn about a low sulfur diet in patients with Crohn's disease. Study participants will be randomized to receive a low sulfur diet or usual diet for 8 weeks. Participants will work with study nutritionists and receive dietary educational materials. Participants will attend 2 in-person visits as well as 6 phone visits during the study. In addition, subjects will undergo testing, including a test to measure rectal sensation, a test to look for small intestinal bacterial overgrowth, and a test to measure leaky gut.

DETAILED DESCRIPTION:
Even in the absence of active inflammation, persistent symptoms are reported in up to 46% of inflammatory bowel disease (IBD) patients, especially in Crohn's disease (CD). While persistent symptoms in quiescent Crohn's disease result in worsened quality of life and worse outcomes, evidence-based treatments do not currently exist due to lack of mechanistic understanding of this condition. The gut microbiome, which are the microbes that live in our gut, have been suggested as a potential cause of persistent symptoms. Diet is a major influence on the microbiome and may have a modifiable impact on persistent symptoms in Crohn's disease. However, this has not been well established.

The investigators propose a study period of approximately 8 weeks to evaluate the effects of a low sulfur diet in Crohn's disease. Participants will have an initial phone visit to determine eligibility to participate in the study and to review potential participants normal diet with a study nutritionist.

The treatment phase of 8 weeks will begin at the baseline visit (week 0). Participants will be randomized to receive a low sulfur diet or usual diet for 8 weeks. Participants on the low sulfur diet will meet with the study nutritionist to receive educational materials and recipes for the low sulfur diet. During this visit, participants will undergo testing, including a rectal barostat test to evaluate rectal sensation, glucose hydrogen breath test to assess for small intestinal bacterial overgrowth, lactulose-mannitol test to evaluate intestinal permeability, and a 24-hour urine sample to measure urine sulfate levels. Participants will be asked to collect saliva, serum, and stool samples.

Participants will then have phone visits every 2 weeks (week 2, week, 4, and week 6). Study nutritionists will monitor their dietary history and answer questions about the low sulfur diet if applicable.

At the conclusion of the 8 weeks, participants will have a final in-person study visit where rectal barostat, glucose hydrogen breath test, lactulose mannitol testing, and 24-hour urine sulfate level will be repeated. Stool and serum samples will be collected by participants.

Optional Low Sulfur Diet for participants randomized to the usual diet:

At the conclusion of the study (week 8), if participants randomized to usual diet are interested, will be offered treatment with a low sulfur diet for the next 8 weeks. Participants will meet with the study nutritionist that will provide educational materials on a low sulfur diet. Participants will have phone visits every 2 weeks (week 10, week 12, and week 14) to review dietary history and answer questions about the low sulfur diet. At the conclusion of the 16 weeks, participants will have a final in-person study visit where they will undergo testing, including a rectal barostat test to evaluate rectal sensation, glucose hydrogen breath test to assess for small intestinal bacterial overgrowth, lactulose-mannitol test to evaluate intestinal permeability, and a 24-hour urine sample to measure urine sulfate levels. Participants will be asked to collect saliva, serum, and stool samples.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of Crohn's disease based on endoscopic, radiographic, and/or histologic findings
* Quiescent Crohn's disease as defined by fecal calprotectin level less than 150 micrograms/gram (mcg/g) stool and/or absence of inflammation on colonoscopy within 30 and 90 days, respectively, of enrollment
* Persistent symptoms will be defined by abdominal pain and/or diarrhea T-scores greater than or equal to 55 by the National Institutes of Health (NIH) Patient-Reported outcomes measurement information system Gastrointestinal scale (PROMIS-GI)

Exclusion Criteria:

* Prior total colectomy
* Presence of an end ileostomy or colostomy in place
* Changes in immunosuppressive medications within the past 4 weeks
* Use of antibiotics or probiotics within the past 4 weeks
* Active or suspected stricture/stenosis of the GI tract
* Habitual vegetarian or vegan diet
* Active or suspected gastrointestinal stricture or stenosis
* Unable or unwilling to follow a low sulfur diet
* Patients who are underweight as defined by BMI < 18.5 kg/m2 or have significant unintentional weight loss as defined by >7.5% body weight in the past 3 months
* Currently pregnant, breastfeeding, and/or unwillingness/inability to use contraception start of the study until the last 13C-mannitol:lactulose test is complete. Sexually active male participants and/or their female partners of reproductive potential must agree to use effective contraception from the start of the study and until the last 13C-mannitol:lactulose test is complete. Women who are breastfeeding must stop breastfeeding during and for at least 12 hours after consuming the 13C-mannitol:lactulose test. Breastfeeding women must pump and dispose of the breastmilk during this time period
* Subjects must agree to not donate sperm or ova (eggs) or breast milk from the start of the study until the last 13C-mannitol:lactulose test is complete.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Dietary Protein Intake for both groups as assessed by 24 hour diet recall | 8 weeks
  Dietary protein intake (animal-based) as assessed by 24 hour diet recall
Dietary Protein Intake as assessed by 24 hour diet recall | Approximately 16 weeks
  Dietary protein intake (animal-based) as assessed by 24 hour diet recall. This is for the group that voluntarily goes on the low sulfur diet after standard of care arm is completed.
Change in 24 hour urinary sulfate | 8 weeks
  Change in 24 hour urinary sulfate level from baseline
Change in 24 hour urinary sulfate | Approximately 16 weeks
  Change in 24 hour urinary sulfate level from baseline. This is for the group that voluntarily goes on the low sulfur diet after standard of care arm is completed

SECONDARY OUTCOMES:
Tolerability of Low Sulfur Diet based on the Visual Analog Scale (VAS) | Week 4
  The VAS has 5 questions in which participants are asked about knowledge, purchase, preparation, ease of following the diet, and overall tolerability of the sulfur diet. Each question participants will score between 0-100 (higher score is more tolerable with total points of 500).
Tolerability of Low Sulfur Diet based on the Visual Analog Scale (VAS) | Approximately week 12
  The VAS has 5 questions in which participants are asked about knowledge, purchase, preparation, ease of following the diet, and overall tolerability of the sulfur diet. Each question participants will score between 0-100 (higher score is more tolerable with total points of 500). This is for the group that voluntarily goes on the low sulfur diet after standard of care arm is completed.
Tolerability of Low Sulfur Diet based on the Visual Analog Scale (VAS) | Week 8
  The VAS has 5 questions in which participants are asked about knowledge, purchase, preparation, ease of following the diet, and overall tolerability of the sulfur diet. Each question participants will score between 0-100 (higher score is more tolerable with total points of 500).
Tolerability of Low Sulfur Diet based on the Visual Analog Scale (VAS) | Approximately 16 weeks
  The VAS has 5 questions in which participants are asked about knowledge, purchase, preparation, ease of following the diet, and overall tolerability of the sulfur diet. Each question participants will score between 0-100 (higher score is more tolerable with total points of 500). This is for the group that voluntarily goes on the low sulfur diet after standard of care arm is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Lee, MD, MS, Principal Investigator — Assistant Professor
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
To be determined